CLINICAL TRIAL: NCT04903990
Title: Fetal Microchimerism and Fetal Stem Cells in Breast Cancer: Analysis of Circulating Fetal Cell Sub-populations in Women With Breast Cancer. CIRCULATING FETAL CELLS AND BREAST CANCER
Brief Title: Circulating Fetal Cells and Breast Cancer
Acronym: MoSaiC2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ruban Rose (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP190505; 2019-A00703-54 (Other: ID-RCB)
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Microchimerism; Hematopietic fetal cells
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for quantification and characterization of fetal blood stem cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: women 18-50 years
  * with previous history of a male birth
  * scheduled for malignant breast tumor surgery
  Interventions: Other: Blood sample
- Controls: women 18-50 years
  * with previous history of a male birth
  * scheduled for benign breast tumor surgery
  * or cancer free
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — As part of the treatment, 2 EDTA tubes of 10mL will be taken during a scheduled venipuncture as part of the preoperative assessment.

SUMMARY:
After pregnancy, fetal cells remain in a woman's body for years. These cells may be involved in different physiological situations (e.g. wound healing) and diseases (e.g. cancer).The study will evaluate the level of circulating fetal immune cells in patients with breast cancer vs controls with benign breast tumors, and further characterize these fetal cells. Patients participation will be limited to accepting that an additional blood sample is collected on the day of their preop consultation and blood test.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in the female population. The protective mechanism associated with pregnancy is not fully understood.

During pregnancy fetal cells cross the placental barrier and may remain in the maternal circulation even for up to 30 years after childbirth. This phenomenon is called fetal microchimerism.

The presence of circulating fetal cells would have a protective role against breast cancer. However, their phenotype and role in the anti-tumor response is not explored.

The objective of the study is to identify the sub-population (s) of circulating fetal immune cells that may have an impact on the processes of carcinogenesis in breast cancer, in the context of fetal microchimerism.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-50
* having had a male child
* informed and not having objected to participating in the research.

Patients:

- having a diagnosis of breast cancer

Controls:

* operated on for benign breast tumors
* cancer free

Exclusion Criteria:

* autoimmune disease
* immunomodulatory treatment
* history of cancer other than breast cancer
* ongoing hormonal treatment
* women not affiliated to the social security
* under AME (state medical aid)
* under tutorship / curatorship

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: The study population includes only women who have had a male child, premenopausal, aged 18-50 years, who are operated on for breast cancer or who have just been diagnosed with breast cancer.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Percentages of fetal cells in each immune cell subpopulation. | 3 years
  Using fluorescence activated cell sorting method.

SECONDARY OUTCOMES:
Activation markers. | 3 years
  Using immunocytochemistry method.
Cytotoxicity markers. | 3 years
  Using immunocytochemistry method.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie CHABBERT-BUFFET, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital de Tenon-Service de Gynécologie Obstétrique et Médecine de la Reproduction, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided